CLINICAL TRIAL: NCT05005780
Title: Stroke Therapy With Brain Oscillation Synchronized Stimulation: Randomized Controlled Pilot Study to Compare the Therapeutic Effectiveness of a Personalized EEG-triggered Repetitive High-frequency TMS Therapy Protocol With Standard Low-frequency TMS Therapy Protocol in Patients With Spastic Paresis
Brief Title: Stroke Therapy With Brain Oscillation Synchronized Stimulation
Acronym: STROKEBOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07, Version 4
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2021-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- µ-alpha oscillation coupled ipsilesional 100 Hz triplet bursts (Experimental): µ-rhythm (The µ rhythm frequency band is defined by activity falling between 8 and 13 Hz and recorded by scalp electrodes over the sensorimotor cortex during waking neural activity) negative peak triggered TMS of ipsilesional primary motor cortex, consisting of 400 triple pulses at 100 Hz, delivered at a mean inter-triple pulse interval of 3.0 s. Stimulation intensity: 100% resting motor threshold.
  Interventions: Device: Negative peak triggered 100 Hz triplet burst TMS
- contralesional 1 Hz rTMS (Active Comparator): 1200 stimuli to the contralesional primary motor cortex at 1 Hz. Stimulation intensity: 115% resting motor threshold.
  Interventions: Device: 1 Hz rTMS

INTERVENTIONS:
Device: Negative peak triggered 100 Hz triplet burst TMS — MagVenture MagPro X100: Ipsilesional negative peak triggered 100 Hz triplet burst TMS.
  Arms: µ-alpha oscillation coupled ipsilesional 100 Hz triplet bursts
Device: 1 Hz rTMS — MagVenture MagPro X100: Contralesional 1 Hz rTMS.
  Arms: contralesional 1 Hz rTMS

SUMMARY:
This randomized, controlled, double-blind clinical pilot trial investigates the therapeutic potential of a novel personalized therapeutic brain-stimulation protocol in chronic stroke patients with spasticity. Stroke patients will either receive ipsilesional 100 Hz transcranial magnetic stimulation (TMS) triplet burst protocol synchronized to the ongoing µ-alpha oscillation or contralesional 1 Hz repetitive TMS (rTMS) protocol. Motor recovery is assessed directly after as well as three months after completion of the therapy.

DETAILED DESCRIPTION:
Stroke is one of the leading cause for long-term disability worldwide. The standard approach to treat deficits after stroke is a rehabilitation therapy, that follows the stroke event directly. This therapy mainly includes physiotherapy and occupational therapy. Yet, despite intensive rehabilitation efforts, more than half of all stroke patients remain greatly disabled.

Repetitive TMS is capable of inducing plasticity-like effects in the brain, that are expected to enhance adaptive plasticity processes leading to functional regain after stroke. In the motor cortex, brain oscillation-synchronized TMS, i.e. TMS triggered dependent on the phase of instantaneous µ-alpha oscillations as detected by real-time EEG (electroencephalography) analysis, has been shown to consistently increase motor cortical excitability and plasticity effects. We therefore hypothesis that a greater therapeutic potential of TMS to modulate dysfunctional brain networks can be exploited by personalizing TMS therapy to individual brain states (i.e. brain oscillations).

This study aims to investigate the effectiveness of an ipsilesional 100 Hz TMS triplet burst protocol synchronized to the ongoing µ-alpha oscillation compared to the current TMS standard therapy of contralesional 1 Hz rTMS in chronic stroke patients. Both groups will undergo stimulation therapy three times a week, with each session directly followed by physiotherapy. Motor recovery will be assessed directly after as well as three months after completion of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are between 18 to 85 years old
2. Patient suffers from chronic stroke including hand/arm paresis and spasticity
3. Ipsilesional motor evoked potentials (MEPs) can be evoked (EMG > 50uV)
4. RMT of contralesional side < 70% maximum stimulator output (MSO)
5. Patient is willing to comply with the study restrictions.
6. Subject FMA-UE at the lesioned side is <= 60.

Exclusion Criteria

1. Patient is under the age of legal consent.
2. Patient has a history of seizure disorder.
3. Patient with intake of pro-convulsive medication, e.g. , chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, MDMA (ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline, in accord with present consensus guidelines on safety, ethical considerations, and application of TMS in clinical practice and research (Rossi et al., 2009, 2021).
4. Subject with intake of muscle-relaxing medication (e.g. baclofen, tizanidine, gabapentin,tolperisone, THC and derivates)
5. When spasticity is treated with botox there have to be at least tree months since the last injection
6. Patient has a cardiac pacemaker, implanted medication pump, intracardiac line, that is located close to (≤ 10 cm) to the location of activation of the TMS coil or acute, unstable cardiac disease.
7. Patient has an intracranial implant (e.g., aneurysm clips, shunts, stimula-tors, cochlear implants, or electrodes) or any other metal object that is located close to (≤ 10 cm) to the location of activation of the TMS coil (excluding the mouth) and that cannot be safely removed.
8. Patient has participated in another study within 2 weeks prior to the first study visit.
9. Patient is pregnant or trying to get pregnant.
10. Patient is unable to give informed consent.
11. Patient is unable to understand the instructions of the FMA-UE or not motivated to follow these instructions.
12. Patients who have contractions and therefore can't move.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment Upper Extremity (FMA-UE) | Difference of score directly before intervention and score directly after intervention
  Upper limb, affected side
Change in Fugl-Meyer Assessment Upper Extremity (FMA-UE) | Difference of score directly before intervention and score 3 months after intervention
  Upper limb, affected side

SECONDARY OUTCOMES:
Change in Wolf-Motor Function Test | Difference of score directly before intervention and score directly after intervention
  Upper limb, affected side
Change in Modified Ashworth Scale | Difference of score directly before intervention and score directly after intervention
  Upper limb, affected side
Change in PSAD spasticity assessment device score | Difference of score directly before intervention and score directly after intervention
  Upper limb, affected side
Change in Resting-motor-threshold (RMT) | Difference of score directly before intervention and score directly after intervention
  Hand knob, affected hemisphere

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Ziemann, Prof. Dr., Principal Investigator — University Hospital Tübingen, Department of Neurology and Stroke
Locations (1):
- University Hospital Tübingen, Department for Neurology and Stroke, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mahmoud W, Baur D, Zrenner B, Brancaccio A, Belardinelli P, Ramos-Murguialday A, Zrenner C, Ziemann U. Brain state-dependent repetitive transcranial magnetic stimulation for motor stroke rehabilitation: a proof of concept randomized controlled trial. Front Neurol. 2024 Aug 26;15:1427198. doi: 10.3389/fneur.2024.1427198. eCollection 2024. PMID 39253360